CLINICAL TRIAL: NCT01967420
Title: Using Computerised Training to Improve Cognition and Functioning in the First Episode of Psychosis
Brief Title: Cognitive Remediation for First Episode of Psychosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Emily Revell, Postgraduate Researcher, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/NW/0385
Record Dates: First submitted 2013-10-14; First posted 2013-10-22 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Psychosis
Keywords: Cognitive remediation; Social cognition training; First episode psychosis; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Cognitive Remediation; Gene Regulatory Networks; Cognitive Training

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- Cognitive remediation plus social cognition training (Experimental): A combined intervention of 60 minutes of computerised cognitive remediation and 30 minutes of computerised social cognition training.
  Interventions: Behavioral: Cognitive remediation; Behavioral: Social cognition training
- Cognitive remediation alone (Active Comparator): An active control condition consisting of 60 minutes of computerised cognitive remediation and 30 minutes of free computer time.
  Interventions: Behavioral: Cognitive remediation

INTERVENTIONS:
Behavioral: Cognitive remediation — CIRCuiTS is a computerised cognitive remediation program which consists of tasks to improve cognition, the use of strategy training and the teaching of generalisable community functioning skills.
  Other Names: CIRCuiTS; cognitive training
Behavioral: Social cognition training — The social cognition training is a computerised program which aims to improve emotion recognition through a variety of lessons and games.
  Other Names: Mind reading - an interactive guide to emotions
  Arms: Cognitive remediation plus social cognition training

SUMMARY:
This study aims to look at the effectiveness of a combination of cognitive remediation and social cognition training to improve cognition and functioning when compared to cognitive remediation alone. The target population will be those who are experiencing their first episode of psychosis.

DETAILED DESCRIPTION:
A first episode of psychosis is defined as the first experience of positive symptoms, such as hallucinations and delusions, and the behaviour that accompanies it. This is associated with problems in many areas of cognition; the ability to acquire knowledge and understanding. These cognitive symptoms have been found to have a large impact on daily functioning (e.g. accessing education or employment and maintaining relationships) and cannot effectively be treated with medication. Cognitive remediation (CR) is a therapy that aims to improve cognition and, through generalisation of this, improve daily functioning and quality of life. Although it is an area of deficit, social cognition, the ability to perceive and understand emotional states, is often not targeted in cognitive remediation. However, interventions which have focused on providing social cognition training (SCT) alongside CR have shown large improvements in daily functioning.

This study aims to look at the effectiveness of a combination of CR and SCT to improve cognition and functioning when compared to CR alone. The target population will be those who are experiencing their first episode of psychosis. Participants will be recruited from an Early Intervention in Psychosis service which is an NHS service set up to provide rapid treatment for those experiencing psychosis.

Participants will take part in a ten week CR or CR+SCT intervention which will consist of spending 90 minutes a week in a small group setting working through a series of computer games which aim to improve cognition. Interviews and questionnaires regarding daily functioning, cognition, quality of life and symptoms will be used before and after the intervention. Participants will be asked to attend follow-up interviews 6 months after the intervention has ended to complete the measures again to see if any beneficial effects have lasted.

ELIGIBILITY:
Inclusion Criteria:

* Non-affective psychosis
* Premorbid IQ of over 70
* A service user of the early intervention service
* Aged 18 or over (up to the age of 35 which is the limit for the early intervention service)
* Psychiatrically stable enough to attend to completion (no hospitalisations or medication changes in last 4 weeks)

Exclusion Criteria:

* Active substance dependency
* History of severe head injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Emotion Recognition Task | 10 weeks
  The emotion recognition task of the computerised Cambridge neuropsychological test automated battery (CANTAB).

SECONDARY OUTCOMES:
CANTAB schizophrenia battery | 10 weeks and 6 month follow-up
  Additional computerised neuropsychological tests from the CANTAB schizophrenia battery will be used. These are the rapid visual information processing task (RVP), the spatial working memory task (SWM), the paired associates learning task (PAL), one touch stockings of Cambridge task (OTS) and the intra-extra dimensional set shift task (IED).
Specific levels of functioning scale (SLOF) | 10 weeks and 6 month follow-up
  SLOF is an observer-rated set of 6 domains of functioning where ratings are made on 5-point Likert scales based on how often a particular behaviour occurs or how much help is required to perform certain tasks. The 6 domains are: physical functioning, personal care skills, interpersonal relationships, social acceptability, activities and work skills, the final four of which will be used in this study. This will be completed with the participant's primary care team and verified with the participant.
Personal and Social Performance Scale (PSP) | 10 weeks and 6 month follow-up
  An additional measure of functioning, the PSP will be added on to the end of the SLOF. The PSP addresses 4 domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviours. It is scored on a 1-100 scale. This is a validated and reliable measure of functioning with high test-retest reliability. It will be completed by a member of the participant's care team.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Beetschen, Principal Investigator — University of Manchester
Locations (1):
- Bradford Early Intervention in Psychosis Service, Bradford, West Yorkshire, United Kingdom